CLINICAL TRIAL: NCT00682773
Title: Enhancing the Safety of Warfarin in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Qualidigm (Industry)
Responsible Party: Jerry Gurwitz, MD, Executive Director, Meyers Primary Care Institute/University of Massachusetts Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12214; 5R01HS016463 (AHRQ)
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Adverse Drug Events (ADEs)
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Usual care, no educational intervention.
- 2 (Experimental): Usual care, nursing home nursing staff receive educational intervention on effective communication regarding warfarin treatment/care; use of SBAR communication forms.
  Interventions: Other: SBAR

INTERVENTIONS:
Other: SBAR — Educational intervention for nursing staff on effective communication regarding warfarin treatment/care; use of SBAR communication forms.
  Arms: 2

SUMMARY:
Oral anticoagulant therapy with warfarin is essential for the prevention of strokes and other thromboembolic events related to various medical conditions; however, use of this therapy can be associated with an increased risk of serious bleeding. In a previous AHRQ-funded study, we have demonstrated that the prevalence of conditions for which warfarin is indicated is high among frail elderly nursing homes residents, use of warfarin in this setting is very common, and the quality and safety with which warfarin is used is far from optimal. The research described in this application resonates with AHRQ's stated priorities for FY2006. The premise underlying the proposed intervention study is that errors in prescribing and monitoring warfarin for nursing home residents are related more to problems in the system of care, than to deficits in the knowledge base of health care providers. We propose a low technology intervention for improving the quality and safety of anticoagulant therapy with warfarin in the nursing home setting. The intervention focuses on maximizing the effectiveness of communication between the nursing staff and physicians of nursing home residents on warfarin. The intervention will build on an established approach for situation briefing drawn from the U.S. armed forces: SBAR - Situation, Background, Assessment, Recommendation. We will test the effectiveness of this approach through a matched, cluster-randomized trial, with randomization at the level of the nursing home. Our study has the following specific aims: (1) to determine whether a nursing home warfarin management protocol emphasizing facilitated communication to physicians will improve the quality of anticoagulation management, which will be assessed using widely accepted quality measures; (2) to determine whether the intervention will lower the rates of adverse events (bleeds and thromboembolic events) among warfarin-treated residents of intervention group nursing homes compared to control nursing homes; and (3) to produce a toolkit for use by nursing homes that will allow dissemination of this approach to enhancing the quality and safety of warfarin for the frail elderly. If successful, this approach may serve as a model for improving the safety of other medication categories associated with high rates of preventable adverse drug events, and for protecting nursing home residents, and frail elderly cared for in other settings, who are at special risk for medication-related problems.

DETAILED DESCRIPTION:
A. SPECIFIC AIMS Long-term oral anticoagulant therapy with warfarin is essential for the prevention of strokes and other thromboembolic events related to various medical conditions that increase in prevalence in older persons. However, the desire to initiate anticoagulant therapy in an older patient is tempered by concerns about the risk of bleeding. The residents of nursing homes are among the most frail patients in the geriatric population and are at increased risk for drug-related iatrogenic injury not only because of the physiologic declines and pharmacologic changes that occur with aging, but also because of the special clinical and social circumstances that characterize this setting of care for more than 1.7 million Americans who reside in an estimated 16,000 nursing homes across the United States.

We have previously shown that the prevalence of conditions for which warfarin is indicated among nursing home residents is high, use of warfarin among this population is common, and the quality of management of this therapy is suboptimal. As many as 12% of nursing home residents receive warfarin for various reasons (nearly 200,000 nursing home residents nationwide). While oral direct thrombin inhibitors have held some promise as less complicated anticoagulants, ximelagatran has been associated with hepatotoxicity and has not yet received approval by the Food and Drug Administration for use in the U.S. For the foreseeable future, warfarin remains the sole oral anticoagulant available for long-term use in the elderly.

Our prior research conducted under the auspices of an AHRQ-funded Center of Excellence for Patient Safety Research and Practice (PO1HS11534) demonstrated overwhelming evidence of safety problems with warfarin therapy in the nursing home setting. Based on that work, we conservatively estimate that there may be as many as 34,000 fatal, life-threatening, or serious adverse warfarin-related events per year in the nursing home setting, the majority of which may be preventable. These include both bleeds and thromboembolic events. Errors in warfarin prescribing and monitoring are responsible for nearly all of the preventable events; inadequate communication of information regarding prior international normalized ratio (INR) values and interacting medications played an important role in many of these events.

The research study described in the current application resonates with AHRQ's mission and the Agency's stated research priorities for FY2006 (NOT-HS-06-032). This research specifically addresses the gaps in care relating to an important medication therapy management issue in a priority population, elderly residents of nursing homes, a population comprised of individuals with multiple medical conditions who are taking multiple medications; the nursing home setting and structure pose special challenges that can subvert efforts to provide high quality, safe, and effective anticoagulation care to a particularly vulnerable population.

The premise underlying the proposed intervention study is that errors in prescribing and monitoring warfarin for nursing home residents are related to problems in the system of care. The system of medication management in the nursing home includes the nursing staff within the facility, and the physicians, laboratories, and pharmacy vendors generally external to the nursing home who interact to provide services to the residents. While an adverse drug event in this setting may be directly linked to a "human error", the root cause may be defined as the defect in the system that permitted such an error to occur. In the case of warfarin therapy management for nursing home residents, an important root cause is poor information flow. One example is a telephone call to a covering physician about a resident with a urinary tract infection without providing crucial information that the resident is taking warfarin. The result may be an order for an antibiotic that interacts with warfarin, leading to an increased risk of a bleeding complication.

Many system-level interventions have been suggested to address the challenges of warfarin therapy management. At the present time, technology-based strategies such as computerized physician order entry with clinical decision support are less amenable to widespread adoption by nursing homes. Other options such as specialized anticoagulation services are logistically difficult to implement and expensive. In addition, our prior research has suggested that such services do not yet have broad acceptance for use in the nursing home setting. Given these limitations, we propose a low technology intervention for improving the safety of anticoagulation in the nursing home. The intervention focuses on maximizing the effectiveness of communication between the nursing staff and physicians of nursing home residents on warfarin. The intervention will build on an established approach for situation briefing drawn from the U.S. armed forces: SBAR - an acronym standing for Situation, Background, Assessment, Recommendation. We will test the effectiveness of this approach and its level of adoption and acceptance through a randomized trial, and will produce and disseminate a toolkit that can be applied in other nursing homes, as well as assisted living and home health settings. If successful, this approach will serve as a model for improving the safety of other medication categories associated with high rates of preventable adverse drug events, and for protecting nursing home residents at special risk for medication-related problems.

We propose a matched, cluster-randomized trial, with randomization at the level of the nursing home, that has the following specific aims:

1. To determine whether a nursing home warfarin management protocol with facilitated communication to physicians will improve the quality of anticoagulation management. Quality of anticoagulation management will be assessed utilizing two principal quality measures:

   1. the proportion of time that nursing home residents receiving warfarin have their international normalized ratios (INRs) within the target therapeutic range; and
   2. the time to next INR measurement after an out-of-range INR.
2. To determine whether a nursing home warfarin management protocol with facilitated communication to physicians will lower the rates of adverse events (bleeds and thromboembolic events) among warfarin-treated residents of intervention group nursing homes compared to control nursing homes.
3. To produce a toolkit for use by nursing homes that will allow dissemination of this approach to enhancing the quality and safety of warfarin in the nursing home setting.

We propose to perform this study in 26 nursing homes in Connecticut. This study takes advantage of the complementary skills and experience of a multidisciplinary research team with expertise in geriatric medicine, geriatric clinical pharmacology, chronic disease epidemiology, effective clinical communication, and gerontological nursing. This study will serve to extend prior collaborative AHRQ-funded research efforts focused on the long-term care setting, between investigators based at the University of Massachusetts Medical School and Qualidigm (formerly the Connecticut Peer Review Organization), a nationally recognized quality improvement organization with close links to nursing homes across the state of Connecticut.

ELIGIBILITY:
Inclusion Criteria:

* Connecticut nursing homes affiliated with Qualidigm

Exclusion Criteria:

* Nursing homes not affiliated with Qualidigm

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The proportion of time that nursing home residents receiving warfarin have their international normalized ratios (INRs) within the target therapeutic range | one year
The time to next INR measurement after an out-of-range INR. | one year
Rates of adverse events (bleeds and thromboembolic events) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jerry H Gurwitz, MD, Principal Investigator — Meyers Primary Care Institute/University of Massachusetts Medical School
Locations (2):
- United States (2):
  - Qualidigm, Middletown, Connecticut
  - Meyers Primary Care Institute, Worcester, Massachusetts

REFERENCES:
- [Derived] Field TS, Tjia J, Mazor KM, Donovan JL, Kanaan AO, Harrold LR, Reed G, Doherty P, Spenard A, Gurwitz JH. Randomized trial of a warfarin communication protocol for nursing homes: an SBAR-based approach. Am J Med. 2011 Feb;124(2):179.e1-7. doi: 10.1016/j.amjmed.2010.09.017. PMID 21295198